CLINICAL TRIAL: NCT05472701
Title: SWAP-MEAT (Study With Appetizing Plant-Food, Meat Eating Alternatives Trial) Athlete
Brief Title: SWAP-MEAT Athlete: Three Diets on Athletic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 59905
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Health Behavior
Keywords: muscular strength; endurance; plant-based diets; meat alternatives; omnivore diets
MeSH Terms: conditions — Health Behavior | interventions — polybutyl methacrylate

STUDY DESIGN:
Intervention Model Description: SWAP-MEAT Athlete is a randomized crossover trial in which 12 recreational runners and 12 recreational resistance trainers are assigned to one of six possible diet orders. Each diet order contains three phases for four weeks each-Animal, Plant-Based Meat Alternatives (PBMA), and Whole Food Plant-Based (WFPB)-in random order.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole Food Plant-Based (WFPB) (Experimental): 2 meals/day of traditional plant proteins (tofu, quinoa, black beans) and minimized intake of processed food, eggs, and dairy
  Interventions: Behavioral: Diet order: WFPB, PBMA, Animal; Behavioral: WFPB, Animal, PBMA; Behavioral: PBMA, WFPB, Animal; Behavioral: PBMA, Animal, WFPB; Behavioral: Animal, WFPB, PBMA; Behavioral: Animal, PBMA, WFPB
- Plant-Based Meat Alternatives (PBMA) (Experimental): 2 servings/day of plant-based meat alternatives (Beyond Beef, Impossible Burger, Gardein Chick'n)
  Interventions: Behavioral: Diet order: WFPB, PBMA, Animal; Behavioral: WFPB, Animal, PBMA; Behavioral: PBMA, WFPB, Animal; Behavioral: PBMA, Animal, WFPB; Behavioral: Animal, WFPB, PBMA; Behavioral: Animal, PBMA, WFPB
- Animal (Experimental): 2 servings/day of traditional meat products (beef burger, pork, chicken)
  Interventions: Behavioral: Diet order: WFPB, PBMA, Animal; Behavioral: WFPB, Animal, PBMA; Behavioral: PBMA, WFPB, Animal; Behavioral: PBMA, Animal, WFPB; Behavioral: Animal, WFPB, PBMA; Behavioral: Animal, PBMA, WFPB

INTERVENTIONS:
Behavioral: Diet order: WFPB, PBMA, Animal — Participants followed the WFPB, PBMA, and Animal diets (in this order) for 4 weeks each.
Behavioral: WFPB, Animal, PBMA — Participants followed the WFPB, Animal, and PBMA diets (in this order) for 4 weeks each.
Behavioral: PBMA, WFPB, Animal — Participants followed the PBMA, WFPB, and Animal diets (in this order) for 4 weeks each.
Behavioral: PBMA, Animal, WFPB — Participants followed the PBMA, Animal, and WFPB diets (in this order) for 4 weeks each.
Behavioral: Animal, WFPB, PBMA — Participants followed the Animal, WFPB, and PBMA diets (in this order) for 4 weeks each.
Behavioral: Animal, PBMA, WFPB — Participants followed the Animal, PBMA, and WFPB diets (in this order) for 4 weeks each.

SUMMARY:
This study aims to investigate the impact of two plant-based diets-whole food plant-based (WFPB) and plant-based meat alternatives (PBMA)-vs. an omnivorous diet (Animal) on endurance and muscular strength in recreational athletes.

DETAILED DESCRIPTION:
Plant-based diets are environmentally sustainable and beneficial for cardiovascular health, but athletes are often concerned that these diets do not contain enough protein to support athletic performance. However, few randomized trials investigating the effect of plant-based vs. omnivorous diets on athletic performance have been conducted. Within this randomized crossover trial, recreational runners and resistance trainers will be assigned to three diets for four weeks each (WFPB, PBMA, and Animal). PMBA is an emerging, modern type of plant-based diet for which the impact on athletic performance has not yet been assessed. Participants will complete athletic fields at baseline and after each diet, and athletic performance on diets and study feasibility in this cohort of recreational athletes will be assessed. The study design was inspired by the original SWAP-MEAT study that investigated cardiovascular risk factors in adults consuming 8-week omnivorous and plant-based meat alternative diets (Crimarco, 2020).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy omnivorous adults between 18 and 35 years of age who report typically consuming at least 1 serving of meat per day and are willing to consume ~2 servings per day of animal meat, plant-based meat alternatives, and whole-food plant proteins.
* Participants will have been consistent recreational runners or weightlifters (3-4 times per week) for at least the prior 1 year, and currently run or lift 3-4 times per week.
* Runners will engage in at least 150 minutes of moderate-to-vigorous aerobic activity or 75 minutes of vigorous activity per week. All participants will have habitually consumed an omnivorous diet for at least months.
* Participants will have self-reported good health and BMI 18.5-30.0.
* Participants must be able to commit to running or resistance training at least 3-4 times per week for the 12 week duration of the study.

Exclusion Criteria:

* Individuals who have participated in any restrictive diet within the last month, have any known nutrient intolerances, have orthopedic limitations, are participating in any other physical activity or diet study;
* Individuals consuming any performance enhancing drugs or medications known to interfere with athletic performance;
* Individuals who have a chronic disease or eating disorder, are currently pregnant or intend to become pregnant in the next three months, or have an intent to compete in any physical activity competition within the next 3 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Cooper 12-Minute Timed Run Test (Runners) | Baseline, Week 4, Week 8, Week 12
  Change from baseline in distance covered on a 12-minute timed run after each diet phase
Composite Machine Strength Index (Resistance Trainers) | Baseline, Week 4, Week 8, Week 12
  Change from baseline in composite machine strength index (sum of 3-rep max chest press, leg press, and lat pull-down) after each diet phase

SECONDARY OUTCOMES:
Estimated VO2 max (Runners) | Baseline, Week 4, Week 8, Week 12
  Change in VO2 max, estimated from training data compiled by Garmin Forerunner 235 after each diet phase
Maximum push-up and pull-up test | Baseline, Week 4, Week 8, Week 12
  Change from baseline in maximum number of repetitions completed of push-up and pull-ups prior to exhaustion after each diet phase
Dietary intake and adherence | Baseline, Week 4, Week 8, Week 12
  a. Nutrient composition of each diet and adherence to diet in servings of protein source consumed per week, via weekly dietary logs
Diet satisfaction | Week 4, Week 8, Week 12
  Score on Food Acceptability Questionnaire, measuring taste, appeal, and overall diet satisfaction, after each diet. We used the "Food Acceptability Questionnaire", with a minimum value of 1 and a maximum value of 7. A higher score indicates better food acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Garnder, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts AK, Busque V, Robinson JL, Landry MJ, Gardner CD. SWAP-MEAT Athlete (study with appetizing plant-food, meat eating alternatives trial) - investigating the impact of three different diets on recreational athletic performance: a randomized crossover trial. Nutr J. 2022 Nov 16;21(1):69. doi: 10.1186/s12937-022-00820-x. PMID 36384651
- See also: Study description and summary of results — https://med.stanford.edu/nutrition/research/completed-studies/SWAPMEAT-athlete.html